CLINICAL TRIAL: NCT06059404
Title: Tailored Occupational Therapy and Registered Dietitian Services for Home-Delivered Meal Clients: A Pilot Randomized Controlled Trial (SixtyPLUS)
Brief Title: Tailoring OT and RD Services for Home-delivered Meal Clients
Acronym: SixtyPLUS
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Ohio State University (Other)
Collaborators: LifeCare Alliance (Unknown)
Responsible Party: Principal Investigator, Lisa Juckett, Principal Investigator, Ohio State University
Allocation: Randomized | Model: Factorial | Masking: Single | Purpose: Treatment
Other Study IDs: 2023H0248
Record Dates: First submitted 2023-09-22; First posted 2023-09-28 (Actual); Last update posted 2025-04-03 (Actual); Status verified 2025-03

CONDITIONS: Diet, Food, and Nutrition; Accidental Fall; Diabetes Mellitus; Heart Diseases
MeSH Terms: conditions — Diabetes Mellitus; Heart Diseases | interventions — Meals

STUDY DESIGN:
Who Masked: Outcomes Assessor
Masking Description: Outcomes assessor will be blinded to participant group assignment
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Meals only (No Intervention): ARM 1: Meals only. Participants randomized to receive "meals only" will receive 14 frozen meals, delivered 1x/week, for 3-months. Participants will be provided with a menu of 40 meal options and instructions for how to select their meals and change weekly meal selections (if desired). Participants in this arm will also receive nutrition education and fall prevention handouts. Nutrition education handouts will indicate which of LifeCare Alliance's meals are considered to be "heart healthy" as well as "diabetic-friendly." Participants will have the autonomy to select their own meals according to their preferences and their ability to self-manage their own health conditions (e.g., diabetes, cardiovascular disease). Fall prevention education handouts will provide guidance on how to reduce fall risk at home and modify the home environment to eliminate fall hazards.
- Meals + registered dietitian services (Active Comparator): ARM 2: Meals + registered dietitian services. Participants randomized to receive "meals + RD only" will receive 14 frozen meals, delivered 1x/week, for 3-months. In addition to receiving nutrition education and fall prevention handouts, participants in this arm will have a telephone-based nutrition assessment completed by one of LifeCare Alliance's registered dietitians who will assign participants a nutrition diagnosis (e.g., overconsumption of carbohydrates) within 60 days of study enrollment.
  Interventions: Behavioral: Meals + RD services only
- Meals + occupational therapy services (Active Comparator): ARM 3: Meals + occupational therapy services. Participants randomized to this arm will receive 14 frozen meals, delivered 1x/week, for 3-months and be able to make weekly meal selections from LifeCare Alliance's full list of 40 meals. In addition to receiving nutrition education and fall prevention handouts, participants in this arm will be contacted (within 30 days of study enrollment) by one of Lifecare Alliance's occupational therapists to complete a phone screen to determine each participant's occupational therapy needs (e.g., home safety/fall risk hazards, need for durable medical equipment).
  Interventions: Behavioral: Meals + OT services only
- Meals + registered dietitian + occupational therapy services (Experimental): ARM 4: Meals + registered dietitian services + occupational therapy services. Participants in this arm will receive 14 frozen meals, delivered 1x/week, for 3-months as well as the same nutrition education and fall prevention handouts as provided in Arms 1-3. Additionally, participants will receive the combination of dietitian and OT services as provided in Arms 2 and 3 and have the same autonomy to make their own weekly meal selections from a curated list provided by the dietitian.
  Interventions: Behavioral: Meals + RD + OT services

INTERVENTIONS:
Behavioral: Meals + RD services only — Registered dietitians (RD) will provide tailored dietitian counseling and nutrition education
  Arms: Meals + registered dietitian services
Behavioral: Meals + OT services only — Occupational therapists (OT) will provide tailored home safety recommendations and fall prevention education/strategies
  Arms: Meals + occupational therapy services
Behavioral: Meals + RD + OT services — A combination of tailored registered dietitian and occupational therapy services will be provided
  Arms: Meals + registered dietitian + occupational therapy services

SUMMARY:
This is a single-blinded, four-arm randomized controlled trial that will compare health outcomes of home-delivered meal clients. The purpose of this pilot study is to explore which service model is most effective for improving nutritional status, disease management, fall risk, and adherence to meal recommendations. Participants will be randomized into one of four study arms: In Arm 1: clients will receive home-delivered meals and basic nutrition education and fall prevention education. In Arm 2: clients will receive home-delivered meals plus dietitian services. In Arm 3: clients will receive home-delivered meals plus occupational therapy services. In Arm 4: clients will receive home-delivered meals plus dietitian and occupational therapy services. Outcomes will be assessed at baseline and at 3-month follow-up.

DETAILED DESCRIPTION:
Participants will be randomized into one of four study arms: ARM 1 - Meals only: Participants randomized to receive "meals only" will receive 14 frozen meals, delivered 1x/week, for 3-months. Participants will be provided with a menu of 40 meal options and instructions for how to select their meals and change weekly meal selections (if desired). Participants in this arm will also receive nutrition education and fall prevention education via standard handouts. Nutrition education handouts will indicate which of LifeCare Alliance's meals are considered to be "heart healthy" as well as "diabetic-friendly." Participants will have the autonomy to select their own meals according to their preferences and their ability to self-manage their own health conditions (e.g., diabetes, cardiovascular disease). Fall prevention education handouts will provide guidance on how to reduce fall risk at home and modify the home environment to eliminate fall hazards. ARM 2 - Meals + registered dietitian services: Participants randomized to receive "meals + RD only" will receive 14 frozen meals, delivered 1x/week, for 3-months. In addition to receiving nutrition education and fall prevention handouts, participants in this arm will have a telephone-based nutrition assessment completed by one of LifeCare Alliance's registered dietitians who will assign participants a nutrition diagnosis (e.g., overconsumption of carbohydrates) within 60 days of study enrollment. During the same phone call, the registered dietitian will also assist participants with their initial meal selections and encourage participants to contact the dietitian with follow-up questions or concerns via phone. Participants will be able to make weekly meal selections based on an approved menu of meals tailored (by a dietitian) to the health needs of the participant. Additionally, dietitians will initiate at least one follow-up phone call no later than 45 days after the nutrition assessment is completed. ARM 3 - Meals + occupational therapy services: Participants randomized to this arm will receive 14 frozen meals, delivered 1x/week, for 3-months and be able to make weekly meal selections from LifeCare Alliance's full list of 40 meals. In addition to receiving nutrition education and fall prevention handouts, participants in this arm will be contacted (within 30 days of study enrollment) by one of Lifecare Alliance's occupational therapists to complete a phone screen to determine each participant's occupational therapy needs (e.g., home safety/fall risk hazards, need for durable medical equipment). Within 30 days after the phone screen, the occupational therapist will then complete an in-home assessment with the participant and provide any initial interventions, equipment, exercises, education as indicated. Within 45 days of the in-home assessment/treatment encounter, the OT will complete an in-home OR phone-based (at the OT's discretion) follow-up session to determine participants' adherence to fall prevention recommendations. All participants randomized to this arm will also be encouraged to call the occupational therapist with questions or concerns over the 3-month study period. ARM 4 - Meals + registered dietitian services + occupational therapy services: Participants in this arm will receive 14 frozen meals, delivered 1x/week, for 3-months as well as the same nutrition education and fall prevention handouts as provided in Arms 1-3. Additionally, participants will receive the combination of dietitian and OT services as provided in Arms 2 and 3 and have the same autonomy to make their own weekly meal selections from a curated list provided by the dietitian.

ELIGIBILITY:
Inclusion Criteria:

1. Self-reported diagnosis of cardiovascular disease (cardiovascular disease may include: hypertension, high cholesterol, congestive heart failure, heart attack or myocardial infarction, peripheral artery disease, stent placement, coronary artery disease, coronary artery bypass graft) or diabetes
2. Over 60 years of age
3. Has one of the following fall risk factors: Uses an assistive mobility device (cane, walker, or wheelchair); Has a fear of falling; Has fallen in the past 12 months; Feels unsteady when standing or walking;
4. Able to store 14 frozen meals/week;
5. Able to reheat meals

Exclusion Criteria:

1. Individuals already receiving home-delivered meals from LifeCare Alliance or other meal agency (within past 6-months)
2. Individuals residing in residential care or a skilled nursing facility

Min Age: 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 56 (Actual)
Dates: Start 2023-09-20 (Actual); Primary Completion 2024-05-29 (Actual); Study Completion 2024-07-31 (Actual)

PRIMARY OUTCOMES:
Mini Nutritional Assessment-Short Form | Baseline and 3-months
  Determine level of malnutrition status

SECONDARY OUTCOMES:
Summary of Diabetes Self-Care Activities Measure | Baseline and 3-months
  Assess management of diabetes as well as heart disease
Falls efficacy scale | Baseline and 3-months
  Assess concerns with falling during daily activities

CONTACTS AND LOCATIONS:
Locations (1):
- LifeCare Alliance, Columbus, Ohio, United States

REFERENCES:
- [Derived] Juckett LA, Joshi S, Hyer JM, Hariharan G, Thomas KS, Sathya TS, Howard ML, Bunck LE, Rowe ML, Devier A, Parrett K; LifeCare Alliance SixtyPLUS Team. Occupational therapy and registered dietitian services to reduce fall risk among home delivered meal clients: a randomized controlled feasibility trial. BMC Geriatr. 2025 May 10;25(1):325. doi: 10.1186/s12877-025-06008-2. PMID 40348980
- [Derived] Juckett LA, Joshi S, Hyer JM, Hariharan G, Thomas KS, Sathya TS, Howard ML, Bunck LE, Rowe ML, Devier A, Parrett K; LifeCare Alliance SixtyPLUS Team. Tailoring registered dietitian and occupational therapy services for home-delivered meal recipients: feasibility study protocol for a randomized controlled trial. Pilot Feasibility Stud. 2025 Apr 5;11(1):41. doi: 10.1186/s40814-025-01623-7. PMID 40188322